CLINICAL TRIAL: NCT07368777
Title: Comparison of Genotype-Based Dietary Counseling Versus Standard Dietary Counseling on Weight Loss and Fat Mass Reduction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Metropolitan College (Other)
Responsible Party: Principal Investigator, Angeliki Kapellou, Principal Investigator, Metropolitan College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 001
Record Dates: First submitted 2026-01-20; First posted 2026-01-27 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Overweight; Overweight and Obesity; Adiposity
Keywords: genotype-based nutrition; dietary counseling; weight loss; nutrigenetics
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genotype-Based Dietary Counseling (Experimental): Participants in this arm will receive dietary counseling tailored according to their genetic profile. Dietary recommendations will be provided by qualified nutrition professionals and will be based on individual genetic information in combination with standard nutritional principles. The counseling will be delivered over the course of the intervention period.
  Interventions: Behavioral: Genotype-Based Dietary Counseling
- Standard Dietary Counseling (Active Comparator): Participants in this arm will receive dietary counseling based on general dietary guidelines and standard nutritional recommendations. Counseling will be provided by qualified nutrition professionals over the course of the intervention period, without the use of genetic information.
  Interventions: Behavioral: Standard Dietary Counseling

INTERVENTIONS:
Behavioral: Genotype-Based Dietary Counseling — This intervention consists of dietary counseling informed by individual genetic information. Nutrition guidance is provided by qualified nutrition professionals and aims to support weight management and reduction of body fat over the intervention period.
  Other Names: Nutrigenetic dietary counseling
  Arms: Genotype-Based Dietary Counseling
Behavioral: Standard Dietary Counseling — This intervention consists of dietary counseling based on general dietary guidelines and standard nutrition recommendations. Counseling is delivered by qualified nutrition professionals without the use of genetic information.
  Other Names: General dietary recommendations
  Arms: Standard Dietary Counseling

SUMMARY:
This study aims to compare the effects of genotype-based dietary counseling with standard dietary counseling based on general recommendations on weight loss and reduction of body fat. Participants will receive individualized dietary guidance either informed by genetic information or based on conventional dietary guidelines. Changes in body weight and body composition will be assessed over the course of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years
* Body mass index (BMI) ≥25 kg/m²
* Greek-speaking (able to read and understand Greek and provide informed consent)
* Willing and able to participate in dietary counseling and study assessments for the duration of the study

Exclusion Criteria:

* Current use of pharmacological treatments for weight loss, including but not limited to GLP-1 receptor agonists, appetite suppressants, or other anti-obesity medications
* Participation in any structured weight-loss intervention or program within the previous 3 months, including commercial weight-loss programs or medically supervised dietary interventions
* Use of medications known to significantly affect body weight or body composition, such as systemic corticosteroids, antipsychotic medications, or medications for thyroid disorders
* Pregnancy or lactation
* Presence of medical conditions that may affect body weight, metabolism, or nutritional status, including untreated thyroid disease, severe gastrointestinal disorders, or endocrine disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in Fat Mass (%) | baseline to end of intervention (12 months)
  Change in whole-body fat mass percentage from baseline to end of the intervention

SECONDARY OUTCOMES:
Change in Body Weight | baseline to end of intervention (12 months)
  Change in body weight from baseline to end of the intervention
Change in Lipid Profile | baseline to end of intervention (12 months)
  Change in fasting lipid profile parameters (e.g., total cholesterol, LDL-C, HDL-C, triglycerides) from baseline to end of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Angeliki Kapellou, PhD, Principal Investigator — Dietetics Department, School of Health Sciences, Metropolitan College
Locations (1):
- Dietetics Department, School of Health Sciences, Metropolitan College, Marousi, Greece

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared outside the research team.